CLINICAL TRIAL: NCT02366611
Title: Pain Control Using Neuromodulation in Patients Undergoing Definitive Chemoradiotherapy for Locally Advanced Head and Neck Cancer
Brief Title: Pain Control Using Neuromodulation in Patients Undergoing Definitive Chemoradiotherapy for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, DMedSc, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM 78942; U036889 (Other: UMichigan)
Record Dates: First submitted 2014-12-02; First posted 2015-02-19 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cancer of Head and Neck
Keywords: Cancer Pain; EEG; fNIRS; tDCS
MeSH Terms: conditions — Head and Neck Neoplasms; Cancer Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) (Experimental): tDCS is a method of non-invasive brain stimulation that is based on the application of a weak direct current to the head that flows between two relatively large electrodes-anode and cathode. tDCS offers a unique analgesic modality of central pain neuromodulation by altering the activity of key sensory and motor cortical structures. Participants in this arm will undergo 20 tDCS sessions, tDCS in clinic and remotely supervised tDCS, and 2mA of transcranial direct current stimulation will be applied for 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Chemoradiotherapy Standard of Care (No Intervention): The control group will consist of patients receiving the Standard of care and no neuromodulation.

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is a non-invasive brain neuromodulatory method that involves sending a weak electrical current to the brain. 2mA of tDCS will be applied for 20 minutes at each session and participants will undergo a total of 20 sessions over a 7-week period.
  Arms: Transcranial Direct Current Stimulation (tDCS)

SUMMARY:
The purpose of this study is to determine if Transcranial Direct Current Stimulation (tDCS) can reduce pain perception associated with the effects of receiving definitive radiation therapy or chemoradiotherapy in head and neck cancer (HNCa) patients.

DETAILED DESCRIPTION:
The goal of this study is to investigate the effectiveness of tDCS as a novel pain relief modality for odynophagia due to mucositis in patients with locally advanced head and neck cancer undergoing definitive radiation therapy or chemoradiotherapy. Participants will be randomized into one of two arms: (1) Treatment: radiation/chemoradiotherapy standard of care + tDCS neuromodulation or (2) Control: radiation/chemoradiotherapy standard of care only.

Patients in the treatment arm will undergo tDCS stimulation on the day of their radiation/chemoradiotherapy appointments, prior to receiving treatment when doing tDCS session in clinic or after to receiving treatment when doing tDCS session at home. This will occur daily (5 days per week) during the second and third weeks of therapy, three times per week during the fourth and fifth weeks, and twice per week during the sixth and seventh weeks.

Patients will also have EEG and fNIRS recordings during the study. This will occur at the pre-study visit, the first stimulation appointment, the third week, the 7th week, and during the follow-up appointments (one-week and one-month).

ELIGIBILITY:
Inclusion Criteria:

* Patients with AJCC stage III-IV head and neck malignancy scheduled for definitive radiation therapy or chemoradiotherapy, and who are capable of understanding and adhering to the protocol requirements.

Exclusion Criteria:

* Substantial dementia
* Patients are actively being treated for another cancer at the time of enrollment.
* Any condition that would prevent use of tDCS including skull abnormality, implanted metal, implanted electronic device, seizure disorder, neurologic condition.
* Use of an investigational drug or device within 30 days of study screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DaSilva, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Started | 10 | 1
Completed | 8 | 1
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care | Total
Number analyzed (Participants) | 10 | 1 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.1) | 58 (NA) — Because only one participant was recruited in this group, therefore no standard deviation was calculated. | 60.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 8 | 1 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: A Visual Analog Scale (VAS) will be used to assess patient-reported odynophagia at weekly Radiation Oncology on-treatment visits (OTVs). The VAS is a traditional pain assessment tool that has been used and validated widely in both clinical and research settings, including studies of oral mucositis pain. This scale ranges from 0-100, in which 0 means no odynophagia, and 100 means highest level of odynophagia ever.
Time Frame: Pre-treatment (baseline), throughout treatment (once a week for 7 weeks), 1 week and 1 month follow-ups (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Number analyzed (Participants) | 7 | 1
score on a scale
  Pre Study | 16 (22) | 2
  Week1 | 11 (14) | 0
  Week2 | 11 (14) | 0
  Week3 | 25 (19) | 0
  Week4 | 34 (31) | 0
  Week5 | 32 (28) | 0
  Week6 | 40 (19) | 0
  Week7 | 36 (18) | 0
  Follow Up Week 1 | 29 (19) | 0
  Follow Up Month 1 | 31 (15) | 0

2. Primary Outcome: EEG Power Spectrum Week1/Week7
Description: EEG data power spectrum analysis. Week1 and Week 7 difference. Note: the control participant's data was not reported due to limited number of participant in the control group. The report was divided into five frequency bands:
  * Delta = 0-4 Hz
  * Theta = 4-7 Hz
  * Alpha = 8-15 Hz
  * Beta= 16-31 Hz
  * Gamma 32-50 Hz
  The data was recorded at P3, Fz, Cz, F3, Fp1, Fp2 points in the international 10-20 system.
  The analysis was done using EEGLab V 14.1.1.
Time Frame: Week1/Week7
Measure: Mean (Standard Deviation); unit: Power(10*log10(muV))^2
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Number analyzed (Participants) | 4 | 1
Power(10*log10(muV))^2
  Delta_Week1_P3 | 118.9 (2.4) | 111
  Theta_Week1_P3 | 115.3 (0.3) | 86.9
  Alpha_Week1_P3 | 115.4 (0.5) | 74
  Beta_Week1_P3 | 114.2 (0.2) | 61.6
  Gamma_Week1_P3 | 115 (0.3) | 50.1
  Delta_Week7_P3 | 129.5 (3.3) | 127.6
  Theta_Week7_P3 | 123.5 (1.5) | 91.7
  Alpha_Week7_P3 | 118.3 (1.8) | 78.9
  Beta_Week7_P3 | 112.0 (2.0) | 66.9
  Gamma_Week7_P3 | 107.4 (1.0) | 55.4
  Delta_Week1_Fz | 118.6 (2.8) | 126.4
  Theta_Week1_Fz | 114.7 (0.2) | 90.5
  Alpha_Week1_Fz | 113.3 (1.4) | 77.5
  Beta_Week1_Fz | 110.8 (0.2) | 64.5
  Gamma_Week1_Fz | 111.7 (0.4) | 51.3
  Delta_Week7_Fz | 146.7 (2.9) | 127.1
  Theta_Week7_Fz | 141.9 (1.6) | 91.2
  Alpha_Week7_Fz | 137.1 (1.7) | 78.6
  Beta_Week7_Fz | 129.3 (2.1) | 68.1
  Gamma_Week7_Fz | 124.0 (1.2) | 57.6
  Delta_Week1_Cz | 117.9 (2.5) | 125.5
  Theta_Week1_Cz | 114.3 (0.2) | 89.6
  Alpha_Week1_Cz | 113.3 (1.3) | 76.5
  Beta_Week1_Cz | 110.7 (0.3) | 63.7
  Gamma_Week1_Cz | 111.4 (0.3) | 51
  Delta_Week7_Cz | 141.7 (3.1) | 126.5
  Theta_Week7_Cz | 136.5 (1.6) | 90.6
  Alpha_Week7_Cz | 132.3 (1.5) | 77.9
  Beta_Week7_Cz | 123.8 (2.5) | 67.1
  Gamma_Week7_Cz | 118.3 (1.1) | 56.4
  Delta_Week1_F3 | 118.6 (3.2) | 125.9
  Theta_Week1_F3 | 114.1 (0.3) | 90
  Alpha_Week1_F3 | 113.1 (1.1) | 77
  Beta_Week1_F3 | 110.7 (0.4) | 64
  Gamma_Week1_F3 | 111.1 (0.3) | 49.8
  Delta_Week7_F3 | 140.3 (3.7) | 129.5
  Theta_Week7_F3 | 133.9 (1.2) | 94.1
  Alpha_Week7_F3 | 127.7 (2.1) | 81.1
  Beta_Week7_F3 | 121.3 (2.1) | 69.4
  Gamma_Week7_F3 | 116.1 (1.2) | 57.2
  Delta_Week1_Fp1 | 119.0 (4.1) | 130
  Theta_Week1_Fp1 | 113.0 (0.5) | 94.1
  Alpha_Week1_Fp1 | 110.9 (1.5) | 81.1
  Beta_Week1_Fp1 | 109.0 (0.2) | 68.3
  Gamma_Week1_Fp1 | 109.0 (0.2) | 53.1
  Delta_Week7_Fp1 | 132.3 (2.9) | 129.5
  Theta_Week7_Fp1 | 127.3 (1.6) | 93.2
  Alpha_Week7_Fp1 | 122.6 (1.5) | 80.3
  Beta_Week7_Fp1 | 114.5 (2.2) | 68.3
  Gamma_Week7_Fp1 | 109.3 (1.1) | 56
  Delta_Week1_Fp2 | 120.4 (3.8) | 128.8
  Theta_Week1_Fp2 | 115.0 (0.5) | 92.9
  Alpha_Week1_Fp2 | 112.4 (1.5) | 80
  Beta_Week1_Fp2 | 108.8 (0.7) | 67.2
  Gamma_Week1_Fp2 | 108.7 (0.2) | 52.6
  Delta_Week7_Fp2 | 129.1 (3.1) | 127.6
  Theta_Week7_Fp2 | 123.0 (1.6) | 91.7
  Alpha_Week7_Fp2 | 119.0 (1.4) | 79
  Beta_Week7_Fp2 | 111.4 (2.1) | 67.9
  Gamma_Week7_Fp2 | 106.6 (1.1) | 56.9

3. Primary Outcome: EEG Spectrum Pre-Post tDCS Session
Description: EEG data power spectrum analysis. Pre/Post-tDCS session. The report was divided into five frequency bands:
  * Delta = 0-4 Hz
  * Theta = 4-7 Hz
  * Alpha = 8-15 Hz
  * Beta= 16-31 Hz
  * Gamma 32-50 Hz
  The data was recorded at P3, Fz, Cz, F3, Fp1, Fp2 points in the international 10-20 system.
  Note: the control participant's data was not reported due to limited number of participant in the control group.
Time Frame: Pre/Post-tDCS Session
Population: Because this piece of result compared EEG data pre- and post- tDCS stimulation, however the control (regular CRT) arm was not stimulated, thus the data were not collected and presented below.
Measure: Mean (Standard Deviation); unit: Power(10*log10(muV))^2
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
Power(10*log10(muV))^2
  Delta_Pre_P3 | 114.8 (2.3)
  Theta_Pre_P3 | 111.0 (0.2)
  Alpha_Pre_P3 | 109.8 (1.1)
  Beta_Pre_P3 | 105.9 (1.0)
  Gamma_Pre_P3 | 104.5 (0.1)
  Delta_Post_P3 | 115.6 (2.6)
  Theta_Post_P3 | 112.2 (0.4)
  Alpha_Post_P3 | 111.9 (1.2)
  Beta_Post_P3 | 109 (0.4)
  Gamma_Post_P3 | 108.8 (0.2)
  Delta_Pre_Fz | 115.4 (2.4)
  Theta_Pre_Fz | 111.4 (0.3)
  Alpha_Pre_Fz | 109.1 (1.5)
  Beta_Pre_Fz | 104.7 (1.1)
  Gamma_Pre_Fz | 103.1 (0.1)
  Delta_Post_Fz | 115.3 (2.6)
  Theta_Post_Fz | 111.7 (0.3)
  Alpha_Post_Fz | 110 (1.6)
  Beta_Post_Fz | 106.7 (0.5)
  Gamma_Post_Fz | 106.3 (0.2)
  Delta_Pre_Cz | 115.9 (2.2)
  Theta_Pre_Cz | 112.1 (0.3)
  Alpha_Pre_Cz | 110 (1.3)
  Beta_Pre_Cz | 105.8 (1.1)
  Gamma_Pre_Cz | 103.9 (0.1)
  Delta_Post_Cz | 116.4 (2.5)
  Theta_Post_Cz | 112.9 (0.2)
  Alpha_Post_Cz | 111.3 (1.4)
  Beta_Post_Cz | 107.4 (0.8)
  Gamma_Post_Cz | 106.5 (0.2)
  Delta_Pre_F3 | 115.7 (2.8)
  Theta_Pre_F3 | 111.4 (0.4)
  Alpha_Pre_F3 | 109.3 (1.2)
  Beta_Pre_F3 | 105.6 (0.8)
  Gamma_Pre_F3 | 104.3 (0.1)
  Delta_Post_F3 | 115.9 (2.8)
  Theta_Post_F3 | 112 (0.2)
  Alpha_Post_F3 | 110.4 (1.4)
  Beta_Post_F3 | 107.8 (0.3)
  Gamma_Post_F3 | 107.6 (0.2)
  Delta_Pre_Fp1 | 115.5 (3.0)
  Theta_Pre_Fp1 | 110.8 (0.4)
  Alpha_Pre_Fp1 | 108.4 (1.4)
  Beta_Pre_Fp1 | 104.6 (0.9)
  Gamma_Pre_Fp1 | 103 (0.1)
  Delta_Post_Fp1 | 114.8 (2.8)
  Theta_Post_Fp1 | 110.9 (0.3)
  Alpha_Post_Fp1 | 109.0 (1.6)
  Beta_Post_Fp1 | 105.7 (0.5)
  Gamma_Post_Fp1 | 105.1 (0.1)
  Delta_Pre_Fp2 | 114.9 (2.7)
  Theta_Pre_Fp2 | 110.4 (0.4)
  Alpha_Pre_Fp2 | 108 (1.5)
  Beta_Pre_Fp2 | 104 (0.9)
  Gamma_Pre_Fp2 | 102.4 (0.1)
  Delta_Post_Fp2 | 114.8 (3.0)
  Theta_Post_Fp2 | 110.7 (0.2)
  Alpha_Post_Fp2 | 108.9 (1.5)
  Beta_Post_Fp2 | 105.9 (0.4)
  Gamma_Post_Fp2 | 105.2 (0.1)

4. Secondary Outcome: Oral-Mucositis Weekly Evaluation - Overall
Description: 1-7 scale grading self-evaluated overall physical condition, 7= Excellent, 1 = Very poor.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Number analyzed (Participants) | 7 | 1
score on a scale
  Pre-Study | 4.9 (1.1) | 7
  Week1 | 5 (1) | 7
  Week2 | 4.8 (1.5) | 7
  Week3 | 4.6 (1.2) | 7
  Week4 | 4.9 (0.6) | 7
  Week5 | 4.7 (0.7) | 7
  Week6 | 4.7 (0.7) | 7
  Week7 | 4.9 (0.8) | 7
  FollowUp-Week1 | 4.5 (1) | 7
  FollowUp-Month1 | 4.6 (0.9) | 7

5. Secondary Outcome: Patient Weight
Description: Participant's weight each measurement time point. Note: 0 means data missing.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pound
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Number analyzed (Participants) | 7 | 1
pound
  Pre-Study | 229.2 (40.6) | 136.5
  Week1 | 224.2 (42.0) | 140
  Week2 | 246.2 (33.2) | 139.3
  Week3 | 221.9 (38.5) | 137.5
  Week4 | 222.8 (41.6) | 140.6
  Week5 | 218.7 (38.4) | 133
  Week6 | 210.7 (37.8) | 132.8
  Week7 | 212.6 (37.6) | 131.9
  FollowUp-Week1 | 220.8 (27.5) | 132
  FollowUp-Month1 | 206.2 (35.5) | 127.9

6. Secondary Outcome: Positive and Negative Affect Schedule
Description: The General Positive and General Negative scores in the PANAS forms are reported for both pre- and post- treatment. The General Positive (GP) and General Negative (GN) scores were reported. Each score ranges from 10-50, in which 10 = lowest (positive/negative emotional level) and 50 = highest (positive/negative emotional level).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Number analyzed (Participants) | 7 | 1
score on a scale
  GP-PRE-PreStudy | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GP-PRE-Week1 | 19 (16) | 37
  GP-PRE-Week2 | 16 (19) | 39
  GP-PRE-Week3 | 11 (19) | 38
  GP-PRE-Week4 | 18 (16) | 39
  GP-PRE-Week5 | 18 (16) | 30
  GP-PRE-Week6 | 23 (13) | 34
  GP-PRE-Week7 | 10 (17) | 37
  GP-PRE-FollowupWeek1 | 21 (15) | 35
  GP-PRE-FollowupMonth1 | 30 (10) | 38
  GN-PRE-PreStudy | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GN-PRE-Week1 | 9 (8) | 13
  GN-PRE-Week2 | 7 (9) | 10
  GN-PRE-Week3 | 4 (8) | 10
  GN-PRE-Week4 | 10 (6) | 10
  GN-PRE-Week5 | 9 (6) | 10
  GN-PRE-Week6 | 11 (5) | 10
  GN-PRE-Week7 | 5 (9) | 10
  GN-PRE-FollowupWeek1 | 10 (7) | 10
  GN-PRE-FollowupMonth1 | 14 (5) | 10
  GP-POST-PreStudy | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GP-POST-Week1 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GP-POST-Week2 | 14 (12) | NA — Data were not collected at the time point.
  GP-POST-Week3 | 14 (14) | NA — Data were not collected at the time point.
  GP-POST-Week4 | 14 (10) | NA — Data were not collected at the time point.
  GP-POST-Week5 | 14 (10) | NA — Data were not collected at the time point.
  GP-POST-Week6 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GP-POST-Week7 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GP-POST-FollowupWeek1 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GP-POST-FollowupMonth1 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GN-POST-PreStudy | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GN-POST-Week1 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GN-POST-Week2 | 13 (12) | NA — Data were not collected at the time point.
  GN-POST-Week3 | 14 (10) | NA — Data were not collected at the time point.
  GN-POST-Week4 | 13 (10) | NA — Data were not collected at the time point.
  GN-POST-Week5 | 14 (10) | NA — Data were not collected at the time point.
  GN-POST-Week6 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GN-POST-Week7 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GN-POST-FollowupWeek1 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.
  GN-POST-FollowupMonth1 | NA (NA) — Data were not collected at the time point. | NA — Data were not collected at the time point.

7. Secondary Outcome: Washington Quality Of Life Questionnaire
Description: The Washington Quality Of Life questionnaire (QOL) is one of the most frequently reported health-related QOL questionnaires in head and neck cancer. This questionnaire scaled from 0 (worst) to 100 (best) according to the hierarchy of response.
Time Frame: Pre-treatment (baseline), Week 7 of treatment, 1 week and 1 month follow-ups (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Number analyzed (Participants) | 7 | 1
score on a scale
  Pre-Study | 18.6 (8.3) | 20
  Week7 | 34.3 (4.9) | 10
  FollowUp-Week1 | 31.7 (6.9) | 10
  FollowUp-Month1 | 28.6 (3.5) | 10

8. Secondary Outcome: Present Pain Intensity Index in McGill Questionnaire Pre-tDCS Treatment
Description: The Present Pain Intensity (PPI) index is recorded as a number ranges from 0 to 5, in which each number is associated with the following words: 0 no pain, 1 mild, 2 discomforting, 3 distressing, 4 horrible, 5 excruciating.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
Number analyzed (Participants) | 7 | 1
score on a scale
  PPI PRE Pre-Study | 0.9 (1.1) | 0
  PPI PRE Week1 | 0.4 (1.0) | 0
  PPI PRE Week2 | 0.7 (1.0) | 0
  PPI PRE Week3 | 1.7 (1.0) | 0
  PPI PRE Week4 | 2.0 (1.4) | 0
  PPI PRE Week5 | 1.8 (1.5) | 0
  PPI PRE Week6 | 1.8 (0.7) | 0
  PPI PRE Week7 | 1.8 (0.9) | 0
  PPI PRE FollowUp Week1 | 1.2 (0.9) | 0
  PPI PRE FollowUp Month1 | 1.7 (0.7) | 0

ADVERSE EVENTS:
Time Frame: 4 years, 11 months
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Chemoradiotherapy Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/1
Other Adverse Events (participants affected / at risk) | 0/10 | 0/1

LIMITATIONS AND CAVEATS:
First, the patient number recruited in the current protocol was small, leading to difficulties in statistics across patients; Second, MRI scanning information did not accompany EEG data for clustering analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT02366611/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT02366611/Prot_SAP_001.pdf